CLINICAL TRIAL: NCT04417088
Title: Assessment of Safety and Feasibility of Exablate Type 2 for Blood-Brain Barrier Disruption (BBBD) With Microbubble Resonators for the Treatment of Recurrent Glioblastoma (rGBM) in Subjects Undergoing Carboplatin Monotherapy
Brief Title: Exablate Blood-Brain Barrier Disruption for the Treatment of rGBM in Subjects Undergoing Carboplatin Monotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT009
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Glioblastoma
Keywords: Exablate; Focused Ultrasound; rGBM
MeSH Terms: conditions — Glioblastoma | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Exablate BBBD with carboplatin (Experimental): Carboplatin will be administered via IV infusion about every 4 weeks for up to 6 cycles. The dosage will be calculated based on subject's creatinine level. On the day of planned carboplatin therapy, subjects will undergo Exablate procedure to open the blood-brain-barrier in the targeted cancerous brain areas prior to Carboplatin administration.
  Interventions: Drug: Carboplatin; Device: Exablate BBBD

INTERVENTIONS:
Drug: Carboplatin — Carboplatin infusion on the day of Exablate BBBD procedure to treat cancerous cells in the brain
Device: Exablate BBBD — BBB opening via Exablate Neuro Type 2 system with microbubble resonators.
  Other Names: Exablate Neuro

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the Exablate Model 4000 Type 2 system when used as a tool to open the blood-brain-barrier (BBB) in subjects with recurrent glioblastoma (rGBM) undergoing carboplatin monotherapy.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, prospective, multi-center, single-arm study to establish the safety and feasibility of blood-brain-barrier disruption (BBBD) combined with intravenous carboplatin for the treatment of rGBM using the Exablate Neuro Model 4000 Type 2 system with microbubble resonators. Adult glioblastoma subjects that are planned for carboplatin chemotherapy will be considered for study enrollment. Eligible subjects will undergo up to 6 cycles of Exablate BBBD procedures in conjunction with carboplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-80 years old
* Histologically confirmed glioblastoma
* Planned for Carboplatin monotherapy
* Be willing and able to provided written informed consent/asent
* Tumor progression after first line chemo radiation
* Recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy
* Women of childbearing potential is confirmed not pregnant. Male and Female subjects utilize highly effective contraception
* Able to communicate verbally

Exclusion Criteria:

* Acute intracranial hemorrhage
* Ferrous metallic implanted objects in the skull or brain
* Prior toxicity with carboplatin chemotherapy
* Women who are pregnant or breastfeeding
* Cerebellar spinal cord or brain stem tumor
* Known active Hepatitis B or Hepatitis C or HIV
* Significant depression not adequately controlled
* Has previously received anti-VEGF or anti-VEGF agents like Avastin
* Cardiac disease or unstable hemodynamics
* Severe hypertension
* History of a bleeding disorder, coagulopathy or with a history of spontaneous tumor hemorrhage
* Active drug or alcohol use disorder
* Known sensitivity to gadolinium-based contrast agents
* Known sensitivity or contraindications to ultrasound contrast agent or perflutren
* Unable to undergo MRI or contraindications to MRI such as non-MRI compatible implanted devices
* Difficulty lying supine and still or severe claustrophobia which cannot be managed with medication
* Severely impaired renal function
* Right to left or bi-directional cardiac shunt
* Cranial or systemic infection requiring antibiotics
* Known additional malignancy that is progression or require active treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 12 months
  All adverse events and/or Serious Adverse Events will be documented and reported according to CTCAE criteria.
Contrast intensity on MR imaging | Immediately after Exablate BBBD procedure
  BBBD will be determined by contrast intensity in sonicated areas on T1 weighted gadolinium-based MR imaging

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio